CLINICAL TRIAL: NCT07265076
Title: Study of Omega-6 Fatty Acids in Patients With Hepatocellular Carcinoma
Brief Title: Role of Omega-6 Fatty Acids in Hepatocellular Carcinoma Development.
Acronym: RO6-HCC
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Maher Sobhy, Resident Doctor of Tropical Medicine and Gastro-enterology, Sohag University
Other Study IDs: 06-HCC-Study-2025-A; Soh-Med--25-10-6MS (Registry Identifier: Medical Research Ethics Committee Faculty of Medicine - Sohag University)
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Hpatocellular
MeSH Terms: conditions — Carcinoma | interventions — Fatty Acids, Omega-6

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC Patients 50-100
- HCC Patients Healthy Controls: HCC Patients: adult patients diagnosed with Hepatocellular carcinoma , meeting inclusion/exclusion criteria healthy controls: age and gender matched healthy adults with no history of liver disease
  Interventions: Dietary Supplement: Omega 6 fatty acid

INTERVENTIONS:
Dietary Supplement: Omega 6 fatty acid — Participants will receive an oral Omega-6 fatty acid dietary supplement in capsule form. The supplement will be administered once daily with meals for a total duration of 8 weeks. Each capsule contains a standardized dose of omega -6 fatty acids, and participants will be instructed to maintain their usual diet during the study period . compliance will be monitored though follow up visits and capsule count . no additional supplements containing omega fatty acids will be allowed during the intervention period .
  Groups: HCC Patients Healthy Controls

SUMMARY:
This observational study investigates the association between serum Omega-6 fatty acids and hepatocellular carcinoma development. Adult HCC patients and age - and gender matched healthy controls will be included. Serum Omega-6 levels will be compared between groups to explore potential correlations with disease presence and severity .

DETAILED DESCRIPTION:
Hepatocellular carcinoma is a leading cause of cancer related deaths worldwide . Omega-6 fatty acids have been suggested to influence liver cancer development .This observational study aims to assess the association between serum Omega-6 fatty acid levels and HCC development .

Adult patients diagnosed with HCC will be recruited from Sohag University Hospital, along with age and gender matched healthy controls . Blood samples will be collected to measure serum Omega-6 levels using standardized bio-chemical assays . clinical and laboratory data , including liver function tests and tumor stage , will also be recorded.

The study will compare Omega-6 levels between HCC patients and controls , and analyze potential correlation with disease severity .Findings may provide insights into the role of Omega-6 fatty acids in HCC pathogenesis and help identify biomarkers for early detection and risk assessment .

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 18 years and above. 2. Patients with hepatocellular carcinoma (confirmed clinically, laboratory, radiologically, or histopathologically).

  3. Ability and willingness to provide informed written consent. 4. For healthy controls: individuals without liver disease or history of malignancy, matched by age and gender.

  5. For cirrhotic controls: patients with liver cirrhosis without evidence of any malignancy, matched by age and gender.

Exclusion Criteria:

1. History of chronic inflammatory (except for liver cirrhosis or HCC) or autoimmune diseases.
2. Current use of omega-6 or omega-3 fatty acid supplements.
3. Presence of other types of cancer.
4. Pregnant or lactating women.
5. presence of severe comorbid condition.

   -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult participants aged 18 years and older will be recruited. The study will include two groups: 1) patients diagnosed with hepatocellular carcinoma confirmed by imaging or histology, and 2) age- and gender-matched healthy controls with no history of liver disease unrelated to HCC, pregnant women, or those currently taking omega fatty acid supplements will be excluded. All participants will provide informed consent prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Serum Omega-6 Fatty Acid Levels | At baseline
  Measurement of circulating levels of Omega-6 fatty acids in blood samples of hepatocellular carcinoma patients and healthy controls using standardized laboratory techniques. The primary outcome will assess the association between serum Omega-6 concentrations and the presence of hepatocellular carcinoma.

REFERENCES:
- See also: General scientific background on hepatocellular carcinoma and related liver diseases — https://pubmed.ncbi.nlm.nih.gov/